CLINICAL TRIAL: NCT01163890
Title: Preventing Mid- and Later-Life Work Limitations: Community-Based Depression Care
Brief Title: Preventing Mid- and Later-Life Work Limitations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: OptumHealth Behavioral Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01AG033125-01A1 (NIH)
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Depression
Keywords: Depression; Work Performance and Productivity; Worksite Intervention
MeSH Terms: conditions — Depression | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WHI (Experimental)
  Interventions: Behavioral: Work and Health Initiative
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Medical or Behavioral Intervention

INTERVENTIONS:
Behavioral: Work and Health Initiative — Telephone-based multi-modal intervention, consisting of: vocational coaching, cognitive-behavioral therapy strategies and care coordination strategies provided by specially-trained EAP counselors
  Arms: WHI
Behavioral: Usual Medical or Behavioral Intervention — Referral to treatment as usual through personal physician, mental health professional, behavioral health program, and/or Employee Assistance Program
  Arms: Usual Care

SUMMARY:
The Work and Health Initiative (WHI) trial is testing an innovative, community-based program that provides mental health and vocational services to workers 50 years or older to improve functioning and reduce productivity loss. The purpose of this study is to test the hypothesis that relative to usual care, the WHI improves the work outcomes of depression and reduces depression-related productivity loss.

DETAILED DESCRIPTION:
National demographic, economic and cultural trends are creating a need for hiring and retaining older workers. However, while many older people will prefer and/or need to work, chronic health problems occurring in mid-life or later can severely disrupt employment. This study will conduct a randomized controlled trial (RCT) of the Work and Health Initiative (WHI). The WHI is an innovative community-based program that provides mental health and vocational services to workers with depression to improve functioning and reduce productivity loss. This study will focus on workers 50 years of age and older. This study will test the hypothesis that relative to usual care, the WHI improves the work outcomes of depression. Study results potentially will result in a new multi-disciplinary method for addressing a serious public health and employment issue.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 45 years
* working ≥ 15 hours/week
* DSM-IV current major depression and/or dysthymia
* Work limitations: at-work productivity loss score ≥ 5%

Exclusion Criteria:

* severe physical health deficits
* non-English speaking or reading
* positive current alcoholism screening
* psychosis
* mania

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
At-work performance deficits and productivity loss as measured by the Work Limitations Questionnaire | 4 months post-randomization
Absenteeism and productivity loss as measured by the Work Limitations Questionnaire Absence Module | 4 months post-randomization

SECONDARY OUTCOMES:
Depression symptom severity as measured by the Patient Health Questionnaire (PHQ-9) | 4 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Debra Lerner, MS, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Adler DA, Lerner D, Visco ZL, Greenhill A, Chang H, Cymerman E, Azocar F, Rogers WH. Improving work outcomes of dysthymia (persistent depressive disorder) in an employed population. Gen Hosp Psychiatry. 2015 Jul-Aug;37(4):352-9. doi: 10.1016/j.genhosppsych.2015.04.001. Epub 2015 Apr 8. PMID 25892151